CLINICAL TRIAL: NCT00561795
Title: A Phase I/II, Open-Label, Multicenter, Two-Arm, Feasibility Study of Pazopanib, Carboplatin, and Paclitaxel in Women With Newly Diagnosed, Previously Untreated, Gynaecological Tumors
Brief Title: Feasibility Study of Pazopanib in Combination With Chemotherapy in Gynaecological Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VEG110190
Record Dates: First submitted 2007-11-19; First posted 2007-11-21 (Estimated); Results first posted 2010-12-07 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2011-03

CONDITIONS: Primary Peritoneal Carcinoma; Tumor; Epithelial Ovarian Cancer; Uterine Disease; Cervix Diseases; Neoplasms, Ovarian; Cancer
Keywords: AGO; Advanced,; Gynaecologic cancer(s),; Genetics; GW786034,; Pazopanib,
MeSH Terms: conditions — Neoplasms; Carcinoma, Ovarian Epithelial; Uterine Diseases; Uterine Cervical Diseases; Ovarian Neoplasms | interventions — pazopanib; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): Oral Pazopanib 800 mg once a day+ carboplatin area under the concentration-time curve (AUC) 5 intravenous (IV) over 1 hour every 3 weeks + paclitaxel 175 mg/m^2 IV over three hours day one q 3 weeks for six cycles
  Interventions: Drug: pazopanib (GW786034); Drug: carboplatin; Drug: paclitaxel
- Arm B (Experimental): Oral Pazopanib 800 mg once a day+ carboplatin AUC 6 IV over 1 hour every 3 weeks + paclitaxel 175 mg/m^2 IV over three hours day one q 3 weeks for six cycles
  Interventions: Drug: pazopanib (GW786034); Drug: carboplatin; Drug: paclitaxel

INTERVENTIONS:
Drug: pazopanib (GW786034) — 800 mg orally once a day for 6 cycles
Drug: carboplatin — IV over one hour every 3 weeks of 6 cycles
Drug: paclitaxel — IV 175 mg/m^2 given over 3 hours on day one of a 21 day cycle for six cycles

SUMMARY:
This is an open-label, two-arm, multicenter feasibility study to evaluate the safety and tolerability of pazopanib in combination with carboplatin and paclitaxel in female subjects with newly diagnosed advanced gynaecological tumors. Subjects will have received no prior therapy for their disease. A minimum of 12 and a maximum of 46 subjects will be enrolled. Dose schemas for each study arm are described in the protocol. For each arm, six subjects will be evaluated in treatment cohorts, which will be expanded to 20 subjects if initial toxicity is acceptable. Overall safety and tolerability of the regimen will be based on dose limiting toxicities, adverse events, and percentage of subjects that complete 6 courses of study treatment. Antitumor activity will be assessed using RECIST criteria and cancer antigen 125 (CA-125) responses.

ELIGIBILITY:
Inclusion criteria:

* Inclusion Criteria
* A subject will be considered eligible for inclusion in this study only if all of the following criteria are met:
* Subjects must provide written informed consent prior to performance of study specific procedures or assessments, and must be willing to comply with treatment and follow up.
* Procedures conducted as a part of routine clinical management of the subject (e.g., blood count, imaging study) and obtained prior to signed informed consent may be utilized for Screening or Baseline purposes provided these tests are obtained as specified in the protocol).
* Female subjects ≥18 years of age with newly diagnosed advanced gynaecological malignancies for whom carboplatin and paclitaxel based chemotherapy is indicated. Patients may have surgery to debulk or resect disease but may not have received chemotherapy or radiotherapy.
* Histological confirmation of the following: epithelial ovarian cancer, endometrial carcinoma, uterine sarcoma, mixed Müllerian tumour, fallopian tube carcinoma, primary peritoneal carcinoma, cervical carcinoma or vulvar carcinoma.
* Performance status must be ECOG 0 1.
* Adequate organ system function as defined in Table 6
* Table 6 Definitions for Adequate Organ Function
* System (Laboratory Values)
* Hematologic:
* Absolute neutrophil count (ANC) (≥ 1.5 X 109/L)
* Hemoglobin1 (≥9 g/dL)
* Platelets (≥100 X 109/L)
* International normalized ratio (INR)(≤ 1.2 X upper limit of normal (ULN))
* Partial thromboplastin time (PTT) (≤1.2 X ULN)
* Hepatic:

p Total bilirubin (≤1.5 X upper limit of normal (ULN))

* AST and ALT (≤ 2.5 X ULN)
* Renal:
* Serum Creatinine (≤ 1.5 mg/dL)
* Or, if serum creatinine >1.5 mg/dL, (≥ 50 mL/min)
* Calculated creatinine clearance
* Urine Protein to Creatinine Ratio2 (<1)
* Patients may not have had a transfusion within 7 days of screening assessment.
* If UPC ≥1, then a 24-hour urine protein must be assessed. Patients must have a 24-hour urine protein value <1g to be eligible.
* Measurable or non-measurable disease.
* A female subject is eligible to enter and participate in the study if she is:
* Of non-childbearing potential (i.e., physiologically incapable of becoming pregnant) including any woman who:
* Has had a hysterectomy, or
* Has had a bilateral oophorectomy (ovariectomy), or
* Has had a bilateral tubal ligation, or
* Is post-menopausal
* Subjects not using hormone replacement therapy (HRT) must have experienced total cessation of menses for ≥ 1 year and be greater than 45 years in age, OR, in questionable cases, have a follicle stimulating hormone (FSH) value >40 mIU/mL and an estradiol value < 40pg/mL (<140 pmol/L).
* Subjects who are using hormone replacement therapy and whose menopausal status is in doubt will be required to use a highly effective method of contraception (as outlined in this inclusion criterion) if they wish to continue their HRT during the study. Otherwise, these subjects must discontinue HRT prior to study enrollment to allow confirmation of post menopausal status. For most forms of HRT, at least 2-4 weeks must elapse between the cessation of HRT and determination of menopausal status; length of this interval depends on the type and dosage of HRT. Following confirmation of post menopausal status, these subjects can resume HRT during the study without use of contraception.
* Childbearing potential, including any female who has had a negative serum pregnancy test within 2 weeks prior to the first dose of study treatment, preferably as close to the first dose as possible, and agrees to use adequate contraception. GSK acceptable contraceptive methods, when used consistently and in accordance with both the product label and the instructions of the physician, are as follow:
* An intrauterine device with a documented failure rate of less than 1% per year.
* Vasectomized partner who is sterile prior to the female subject's entry and is the sole sexual partner for that female.
* Complete abstinence from sexual intercourse for 14 days before exposure to investigational product, through the dosing period, and for at least 21 days after the last dose of investigational product.
* Double-barrier contraception (condom with spermicidal jelly, foam suppository, or film; diaphragm with spermicide; or male condom and diaphragm with spermicide).

Note: Oral contraceptives are not reliable due to potential drug-drug interactions.

* Female subjects who are lactating should discontinue nursing prior to the first dose of study drug and should refrain from nursing throughout the treatment period and for 14 days following the last dose of study drug.
* Recovered from the effects of surgery.
* Prior radiotherapy is permissible, provided at least 4 weeks have elapsed since the last treatment to allow for full bone marrow recovery.

Exclusion Criteria

* A subject will not be eligible for inclusion in this study if any of the following criteria apply:
* Prior use of anticancer therapy (except cytoreductive surgery [debulking]) for their cancer.
* Presence of bulky, residual, squamous cell tumors.
* Is unable to discontinue prohibited medications, as listed in Section 8.2 for 14 days or five half-lives of a drug prior to Visit 1 and for the duration of the study.
* Clinically significant gastrointestinal abnormalities which might interfere with oral dosing, including but not limited to:
* Malabsorption syndrome
* Major resection of the stomach or small bowel that could affect the absorption of study drug
* Active peptic ulcer disease
* Inflammatory bowel disease
* Ulcerative colitis, or other gastrointestinal conditions with increased risk of perforation
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days prior to beginning study treatment.
* Any unstable or serious concurrent condition (e.g., active infection requiring systemic therapy).
* Inadequately controlled hypertension (systolic blood pressure [SBP] of ≥140 mmHg, or diastolic blood pressure [DBP] of ≥ 90 mmHg). Initiation or adjustment of blood pressure medication is permitted prior to study entry provided the subject has 2 consecutive blood pressure readings less than 140/90 mmHg, each separated by a minimum of 24 hours. These readings need to be collected prior to the first dose.
* Hemoptysis within four weeks prior to first dose of study drug.
* Prior major trauma within 14 days prior to first dose of study drug.
* Prior major surgery within 14 days prior to first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer. In the case of surgery involving the bowel, subjects must be 28 days post-surgery to be eligible.
* Prolongation of corrected QT interval (QTc) > 480 msecs.
* History of any one of more of the following cardiovascular conditions within the past 6 months:
* Cardiac angioplasty or stenting
* Myocardial infarction
* Unstable angina
* Symptomatic peripheral vascular disease
* Class III or IV congestive heart failure as defined by the New York Heart Association (NYHA) [See History of cerebrovascular accident (CVA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months.
* Note: Subjects with recent DVT who have been treated with therapeutic anti-coagulant agents (excluding therapeutic warfarin) for at least 6 weeks are eligible.
* Metastatic disease to the brain or leptomeninges.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-09; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- France (2):
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Strasbourg
- Germany (3):
  - GSK Investigational Site, Marburg, Hesse
  - GSK Investigational Site, Wiesbaden, Hesse
  - GSK Investigational Site, Essen, North Rhine-Westphalia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was to occur in Arm B (Arm A6-1 or A6-2) if <2 subjects experienced dose-limiting toxicities (DLTs) while on Arm A5-1 or A5-2. After review of data (pre-specified in protocol) ≥2 subjects in Arms A5-1 and A5-2 experienced DLTs; the study was closed and no subjects were enrolled into Arm B. Three ongoing subjects were taken off regimen.
Groups:
- A5-1: Paclitaxel 175 milligrams (mg)/square meter (m^2) plus carboplatin area under the concentration-time curve (AUC) 5 intravenously (IV) on Day 1 of a 21-day cycle for 6 cycles plus pazopanib 800 mg/day orally starting on Day 1 for the duration of the study
- A5-2: Paclitaxel 175 mg/m^2 plus carboplatin AUC5 intravenously (IV) on Day 1 of a 21-day cycle for 6 cycles plus pazopanib 400 mg/day orally starting on Day 1 for the duration of the study
- A6-1: Paclitaxel 175 mg/m^2 plus carboplatin AUC6 intravenously (IV) on Day 1 of a 21-day cycle for 6 cycles plus pazopanib 800 mg/day orally starting on Day 1 for the duration of the study
- A6-2: Paclitaxel 175 mg/m^2 plus carboplatin AUC6 intravenously (IV) on Day 1 of a 21-day cycle for 6 cycles plus pazopanib 400 mg/day orally starting on Day 1 for the duration of the study
Period: Overall Study
Arm/Group | A5-1 | A5-2 | A6-1 | A6-2
Started | 6 | 6 | 0 | 0
Completed | 2 | 0 | 0 | 0
Not Completed | 4 | 6 | 0 | 0
Not completed — Adverse Event | 3 | 3 | 0 | 0
Not completed — Study Closed/Terminated | 0 | 3 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A5-1 | A5-2 | Total
Number analyzed (Participants) | 6 | 6 | 12
Age Continuous [Mean (Standard Deviation); unit: years] | 55.0 (9.84) | 52.3 (9.85) | 53.7 (9.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White - White/Caucasian/European Heritage | 6 | 6 | 12

OUTCOME MEASURES:

1. Secondary Outcome: Overall Response
Description: Although the study protocol specified several efficacy analyses, due to poor tolerability of the combination regimen and the consequent early withdrawal of most participants, which led to a small sample size, efficacy analyses were not performed. Overall response is defined as the number of participants with CR or PR per Response Evaluation Criteria In Solid Tumors (RECIST): CR, all detectable tumor has disappeared; PR, a >=30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum.
Time Frame: Baseline until either response or progression (up to 2 years)
Measure: Number; unit: participants
Arm/Group | A5-1 | A5-2 | A6-1 | A6-2
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Cancer Antigen (CA-125) Response
Description: Defined as the number of participants who achieved a confirmed CA-125 response, which is defined as at least a 50% reduction in CA-125 levels from a pre-treatment sample.
Time Frame: Baseline until response (up to 2 years)
Measure: Number; unit: participants
Arm/Group | A5-1 | A5-2 | A6-1 | A6-2
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: 18-week Progression Free Survival
Description: Defined as the number participants who have not had radiological disease progression per RECIST, confirmed CA-125 progression, or death due to any cause by the end of 18 weeks.
Time Frame: Baseline to Week 18
Measure: Number; unit: participants
Arm/Group | A5-1 | A5-2 | A6-1 | A6-2
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants Experiencing Serious Adverse Events and Non-serious Adverse Events
Description: Safety and tolerability were measured by the number of participants with serious adverse events and non-serious adverse events. See the "Adverse Event" section of the results record for additional details and data.
Time Frame: Baseline to End of Study (up to a year)
Measure: Number; unit: participants
Arm/Group | A5-1 | A5-2 | A6-1 | A6-2
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Enrollment to End of Study (up to a year)
Arm/Group | A5-1 | A5-2
Serious Adverse Events (participants affected / at risk) | 6/6 | 2/6
Other Adverse Events (participants affected / at risk) | 5/6 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A5-1 (N=6) | A5-2 (N=6)
Neutropenia (Blood and lymphatic system disorders) | 5 | 2
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Ileal Perforation (Gastrointestinal disorders) | 1 | 0
Intestinal Perforation (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Haemoglobin Increase (Investigations) | 0 | 1
Skin Necrosis (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A5-1 (N=6) | A5-2 (N=6)
Abdominal Pain (Gastrointestinal disorders) | 2 | 2
Nausea (Gastrointestinal disorders) | 3 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Vomiting (Gastrointestinal disorders) | 2 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Gastric Disorder (Gastrointestinal disorders) | 1 | 0
Intestinal Perforation (Gastrointestinal disorders) | 1 | 0
Paraesthesia Oral (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 1
Tooth Disorder (Gastrointestinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 3
Acne (Skin and subcutaneous tissue disorders) | 1 | 1
Palmar-Plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Fissures (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 4 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Fatigue (General disorders) | 4 | 3
Mucosal Inflammation (General disorders) | 2 | 0
Pain (General disorders) | 2 | 0
Oedema Peripheral (General disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 0
Catheter Related Infection (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 0 | 2
Urinary Tract Infection (Infections and infestations) | 0 | 1
Headache (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 1
C-Reactive Protein increased (Investigations) | 1 | 0
Haemoglobin Decreased (Investigations) | 1 | 1
Weight Decreased (Investigations) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nervousness (Psychiatric disorders) | 1 | 0
Restlessness (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 0 | 1
Sleep Disorder (Psychiatric disorders) | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
As defined in the protocol, a review of the safety data in Arm A showed that >=2 participants in each regimen of Arm A experienced dose-limiting toxicities. Thus the study was closed to further enrollment and no participants were enrolled into Arm B.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.